CLINICAL TRIAL: NCT04179656
Title: An Open-label, Phase 2 Study of Pyrotinib Maleate in Advanced Solid Tumors Patients With HER2( Erb-B2 Receptor Tyrosine Kinase 2)-Postive
Brief Title: The Basket Study of Pyrotinib Maleate for HER2-Postive Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-HER2
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Solid Tumor; HER2 Gene Mutation; HER-2 Gene Amplification; HER-2 Protein Overexpression
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Treatment (Experimental): This arm for HER2-postive solid tumor
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — 400 mg administered orally, once daily, continuously in 21 day cycles
  Other Names: SHR1258

SUMMARY:
This is an open-label, Phase 2 study exploring the efficacy and safety of 马来酸Pyrotinib Maleate Tablets in patients with solid tumors with activating（harmful） HER2 mutations or with HER2 gene amplification or immunohistochemical staining (IHC) assay showing HER2 is 3+ and / or fluorescence in situ hybridization (FISH) positive.

ELIGIBILITY:
Inclusion Criteria

1. Patients between the ages of 18 and 75;
2. ECOG physical status score 0-2 points;
3. The estimated total survival period is not less than 12 weeks;
4. Patients with HER2-positive solid tumors confirmed by pathology and identified as advanced tumors by clinicians or centers;
5. HER2 positive: refers to standard immunohistochemical staining (IHC) assay showing HER2 is 3+ and / or fluorescence in situ hybridization (FISH) positive or after second generation sequencing shows HER2 amplification and copy number ≥ 3, or There is a HER2 activating mutation identified by the Molecular Oncology Committee (confirmed by the investigator at the test center) ;
6. Imaging studies have at least one measurable lesion with a diameter ≥ 10 mm;
7. Pilotinib has not been used for the past 3 months;
8. The main organs function normally, they meet the following criteria:

   1. Blood routine examination criteria are to comply with:

      ①.Hb≥100 g/L; ②.ANC ≥ 1.5 × 109 / L; ③.PLT≥75×109 /L;
   2. Biochemical tests are subject to the following criteria

      ①.TBIL ≤ 1.5 × ULN (upper limit of normal value);

      ②.ALT and AST ≤ 2.5 × ULN; if there is liver metastasis, ALT and AST ≤ 5 × ULN;

      ③.Serum creatinine ≤ 1.5 × ULN, creatinine clearance ≥ 50ml / min (based on Cockroft and Gault formula);
   3. Heart color ultrasound: Left ventricular ejection fraction (LVEF) ≥ 50%;
9. The patient or his legal guardian understands the test procedure and content and signs an informed consent form (ICF) to provide true and effective information in accordance with the research and follow-up procedures;

Exclusion Criteria:

1. There is a third interstitial fluid that cannot be controlled by drainage or other methods, such as pleural effusion and ascites;
2. It has many factors affecting the oral and absorption of drugs (such as inability to swallow, postoperative gastrointestinal resection, chronic diarrhea and intestinal obstruction);
3. Those who have been confirmed to be allergic to the drug components of this program;
4. Patients who are known to be pregnant or planning to become pregnant, or gestational age patients who are unwilling to take effective contraceptive measures throughout the trial;
5. Patients with severe concomitant diseases or those considered by the investigator to be unsuitable for inclusion.
6. The investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of the study (for administrative reasons or for other reasons).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | at least 3 months
  Objective response rate defined as the patients confirmed complete response or partial response under RECIST 1.0 criteria.

SECONDARY OUTCOMES:
Progression free survival | up to 24 months
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from registration to the earlier of death or disease progression
Duration of Response | up to 24 months
  The first evaluation of treatment efficacy is the time fromcomplete response or partial response to the first assessment of disease progression or death from any cause.
Disease Control Rate | up to 24 months
  Objective response rate defined as the patients confirmed complete response or partial response or stable disease under RECIST 1.0 criteria.
Overall Survival | up to 36 months
  Overall survival estimated using Kaplan-Meier methods is defined as the time from treatment initiation to death by any cause
Safety (Adverse Events and Serious Adverse Events) | up to 36 months
  From consent through 28 days following treatment completion (estimated 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided